CLINICAL TRIAL: NCT01360450
Title: Efficacy of Clonidine in Reducing Iatrogenic-induced Opioid Dependence in Infants:
Brief Title: Clonidine to Treat Iatrogenic-induced Opioid Dependence in Infants
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was treminated because of low accural
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Clonidine NICU-NAS; R21DA029295-01 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2011-05-25 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: opioid withdrawal; Neonatal Pain, Agitation, and Sedation Scale (NPASS); duraclon
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Psychomotor Agitation | interventions — Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Interventions: Infants will receive intravenous or oral clonidine(Duraclon) for the treatment of pain and sedation: Duration: (Clonidine HCL) 1 mcg/kg/dose q4 either iv or po.
  Interventions: Drug: Clonidine HCL
- Control (Placebo Comparator): Intervention: Infants will receive place (saline) (if receiving it IV) or orally (sterile water) if receiving it orally
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Clonidine HCL — At day 5 on opioid and/or benzodiazepine (BZD), the infant will be randomized to receive either placebo (normal saline) or clonidine 1μg/kg/q 4 hrs to a maximum dose of 2μg/kg/q 4. Weaning from the study drug: When the opioid is no longer required, 24 hrs later the study drug (placebo or study drug) will be reduced by 50% and then discontinued 24 hours later provided that the Modified Finnegan scores remain between < 9.
  Other Names: Duraclon
  Arms: Treatment
Drug: saline — Infants randomized to placebo will be administered IV saline or oral sterile water in the same volume as study drug. The placebo will be give every 4 hrs as outlined in the algorithm for the study.
  Other Names: placebo, sterile water, saline
  Arms: Control

SUMMARY:
Thousands of critically ill infants (and children) are exposed to opioids and benzodiazepines to achieve sedation and analgesia as part of routine care in neonatal and pediatric intensive care units. While the use of these agents are undisputedly beneficial in reducing pain and anxiety, improving ventilation, reducing pulmonary vascular resistance and improving outcomes; the consequence is often the development of tolerance and physiologic dependence - similar to prenatal exposure from these same classes of drugs. The investigators have recently reported the results of randomized placebo control trial showing that the addition of clonidine (central alpha 2 agonist) to tapering doses of opioids was efficacious and safe in treating opioid dependence in infants who had moderate to severe neonatal abstinence syndrome from prenatal drug exposure to opioids. Currently, the investigators propose to perform a double-blind, randomized placebo control trial in a cohort of critically ill infants without prenatal drug exposure at Johns Hopkins Hospital to test the overall hypothesis that early addition of clonidine to a cohort of critically ill neonates on mechanical ventilation who are receiving opioids and benzodiazepines for analgesia and sedation will be efficacious and safe in reducing both the incidence and severity of withdrawal symptoms (NICU-NAS); as well as, reducing the time to complete sedative and analgesic drug detoxification. The hypothesis will be tested by addressing 2 specific aims that will determine: 1) the efficacy and safety of clonidine in critically ill infants, and 2) pharmacokinetics and pharmacodynamics using population-based pharmacokinetics in this vulnerable infant population who have only been exposed to these drugs as part of their routine care. Many "standard of care practices" are incorporated in neonatal and pediatric care prior to evidence based studies. This proposal will fill a much needed gap in translating what the investigators have learned about basic mechanisms mediating dependence and withdrawal to proven therapies for vulnerable pediatric populations.

DETAILED DESCRIPTION:
The study will test the following 2 specific aims:

Specific Aim 1

To determine the efficacy and short-term safety of clonidine in reducing the severity of iatrogenic neonatal abstinence syndrome (NAS) by decreasing the time required for complete sedative and analgesic drug detoxification. The investigators will enroll 88 neonates at risk for having moderate to severe NAS in a randomized, double-blinded placebo controlled trial comparing opioid/benzodiazepine administration combined with a placebo (control) vs. opioid/benzodiazepine combined with clonidine. Principal outcome measure will be the difference in length of treatment for complete detoxification. Early safety of clonidine will be determined by monitoring for cardiorespiratory side effects that might be associated with clonidine use in this high risk population.

Specific Aim 2

To determine the pharmacokinetics and pharmacodynamics of clonidine in this critically ill infant population. The investigators will estimate the dose-exposure-response relationship of clonidine in neonates at risk for developing iatrogenic by using nonlinear mixed-effects population pharmacokinetic (PK)-pharmacodynamic (PD) analysis.

ELIGIBILITY:
Inclusion Criteria:

* >35 week Gestational Age (GA) at birth
* <3 months (90 days) old chronological age at the time of enrollment
* Exposed to a minimum five days of continuous narcotic infusion

Exclusion Criteria:

* Neurologic abnormality which would make Neonatal Abstinence Score (NAS) scoring inaccurate
* Major chromosomal abnormality (with the exception of Trisomy 21)
* Infant already enrolled in another randomized, controlled clinical trial

Ages: 5 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estelle B Gauda, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agthe AG, Kim GR, Mathias KB, Hendrix CW, Chavez-Valdez R, Jansson L, Lewis TR, Yaster M, Gauda EB. Clonidine as an adjunct therapy to opioids for neonatal abstinence syndrome: a randomized, controlled trial. Pediatrics. 2009 May;123(5):e849-56. doi: 10.1542/peds.2008-0978. Epub 2009 Apr 27. PMID 19398463
- [Background] Leikin JB, Mackendrick WP, Maloney GE, Rhee JW, Farrell E, Wahl M, Kelly K. Use of clonidine in the prevention and management of neonatal abstinence syndrome. Clin Toxicol (Phila). 2009 Jul;47(6):551-5. doi: 10.1080/15563650902980019. PMID 19566381
- [Background] Pohl-Schickinger A, Lemmer J, Hubler M, Alexi-Meskishvili V, Redlin M, Berger F, Stiller B. Intravenous clonidine infusion in infants after cardiovascular surgery. Paediatr Anaesth. 2008 Mar;18(3):217-22. doi: 10.1111/j.1460-9592.2008.02413.x. PMID 18230064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants recruited from the Neonatal Intensive Unit (NICU) and Pediatric Intensive Unit (PICU) at Johns Hopkins Hospital within 5 days of birth who needed sedation and analgesia as part of treatment.
  Recruitment period was from July 2011 to July 2014. Accrual was very low
Pre-assignment Details: All patients who were enrolled participated in the study.
Groups:
- Treatment: Infants will receive intravenous or oral clonidine(Duraclon) for the treatment of pain and sedation
  Clonidine Hydrochloride: At day 5 on opioid and/or benzodiazepine (BZD), the infant will be randomized to receive either placebo (normal saline) or clonidine 1μg/kg/q 4 hrs to a maximum dose of 2μg/kg/q 4. Weaning from the study drug: When the opioid is no longer required, 24 hrs later the study drug (placebo or study drug) will be reduced by 50% and then discontinued 24 hours later provided that the Modified Finnegan scores remain between < 9.
- Control: Infants will receive place (saline) (if receiving it IV) or orally (sterile water) if receiving it orally
  saline: Infants randomized to placebo will be administered IV saline or oral sterile water in the same volume as study drug. The placebo will be give every 4 hrs as outlined in the algorithm for the study.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 6 | 6
Completed Treatment | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The gestational age of the infant and the birth weight were collected as baseline measurements
Groups:
- Treatment: Infants will receive intravenous or oral clonidine(Duraclon) for the treatment of pain and sedation
  Clonidine HCL: At day 5 on opioid and/or benzodiazepine (BZD), the infant will be randomized to receive either placebo (normal saline) or clonidine 1μg/kg/q 4 hrs to a maximum dose of 2μg/kg/q 4. Weaning from the study drug: When the opioid is no longer required, 24 hrs later the study drug (placebo or study drug) will be reduced by 50% and then discontinued 24 hours later provided that the Modified Finnegan scores remain between < 9.
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Birth Weight [Mean (Standard Deviation); unit: grams] | 3084 (0.59) | 3250 (0.9) | 3160 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Detoxification
Description: Time to complete detoxification is defined as 48 hrs off all opioids/benzodiazepines and study drug with acceptable withdrawal scores of <9 (on average we expect the infant to be enrolled in the study for 2-4 weeks). The scale used to assess withdrawal was the Modified Finnegan Neonatal Withdrawal Scale, which ranges from 0-41, 0 represents no withdrawal and 41 represent maximum withdrawal.
Time Frame: up to 4 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 6 | 6
days
  total days on narcotics | 89.5 (137) | 37.2 (10)
  duration on study drug in days | 21 (18.1) | 14.2 (8.5)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Other; p > 0.05, ANOVA — yes the P value was adjusted for multiple comparisons; 2 sided ANOVA; Mean Difference (Final Values) = 0.05 — Mean difference between the two treatment arms

2. Secondary Outcome: Cardiovascular Side-effects Changes HR and BP
Description: Changes in Heart Rate (HR) and BP for 48 hrs after starting study drug and for 48hrs after stopping study drug
Time Frame: 48 hrs after starting study drug and for 48hrs after stopping study drug
Population: No data is available for this outcome measure, as it was not collected.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cumulative Dose of Opioid and Benzodiazepine
Description: We will determine the total amount of opioid and benzodiazepine needed from the start of detoxification to the end of the the detoxification.
Time Frame: 2-4 weeks
Population: No data is available for this outcome measure, as it was not collected.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No